CLINICAL TRIAL: NCT03110341
Title: Effect of Early Application of Recombinant Human Erythropoietin in Premature Infants on White Matter Lesions and Neurodevelopmental Outcome
Brief Title: Effect of Erythropoietin in Premature Infants on White Matter Lesions and Neurodevelopmental Outcome
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Xian Children's Hospital (Other Government); Shaanxi Provincial People's Hospital (Other); Second Affiliated Hospital of Xi'an Jiaotong University (Other); Tang-Du Hospital (Other); Xijing Hospital (Other); Xi'an No.4 Hospital (Unknown); Northwest Women's and Children's Hospital, Xi'an, Shaanxi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XJTU1AF-CRF-2016-023
Record Dates: First submitted 2017-03-15; First posted 2017-04-12 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Premature Infants; Intracranial Hemorrhages; Periventricular Leukomalacia; Cerebral Palsy
MeSH Terms: conditions — Premature Birth; Intracranial Hemorrhages; Leukomalacia, Periventricular; Cerebral Palsy | interventions — Erythropoietin; epoetin beta; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Erythropoietin (Experimental): Erythropoietin is administered 750U/kg intravenously every other day for 2 weeks (a cumulative dose of 5,250U/kg over the course of 7 separate intravenous injections regardless of gestational age), starting with the first dose within 72 hours after birth. A single dose consisted of 750U EPO per kg of birth weight dissolved in 3mL/kg normal saline was administered intravenously during a period of 5 minutes.
  Interventions: Drug: Normal saline
- Normal saline (Placebo Comparator): Normal saline is administered 3ml/kg intravenously every other day for 2 weeks, starting with the first dose within 72 hours after birth. Similarly, the placebo dose consisted of 3mL of normal saline per kilogram birth weight was administered intravenously during a period of 5 minutes.
  Interventions: Drug: Erythropoietin

INTERVENTIONS:
Drug: Erythropoietin — rhEPO 750U/kg was injected within 72h after birth, subsequent injection was given every other day for 2 weeks (a cumulative dose of 5,250U/kg over the course of 7 separate intravenous injections.
  Other Names: Epoetin Beta
  Arms: Normal saline
Drug: Normal saline — placebo (Normal saline 3 ml/kg birth weight) was injected within 72h after birth, subsequent injection was given every other day for 2 weeks.
  Other Names: NaCl 0.9%
  Arms: Erythropoietin

SUMMARY:
Preterm and very preterm infants are at risk of developing encephalopathy of prematurity and long-term neurodevelopmental delay. Magnetic resonance imaging (MRI) allows the characterization of specific features of encephalopathy of prematurity, including structural changes of brain white matter and gray matter. This study wants to investigate important evidence that early repeated high-dose rhEPO(5250 IU/kg) treatment improves long-term neurological outcomes in very preterm infants and without obvious adverse effects.

DETAILED DESCRIPTION:
HYPOTHESIS Early administration of human erythropoietin (EPO) in preterm infants reduces perinatal injury to the brain and improves neurodevelopmental outcome at 24 months corrected age.

PRIMARY OBJECTIVE To determine whether cerebral outcome is improved if infants born between 28 0/7 and 34 6/7 gestational weeks at birth receive erythropoietin in high dose in the first two weeks after birth.

Biomarkers of encephalopathy of prematurity assessed on magnetic resonance imaging (MRI) at term equivalent age.

RATIONALE Erythropoietin (EPO) was first recognized for its hematopoietic properties; recombinant human EPO (rhEPO) has been used to treat a number of anemic states, including early and late anemia of prematurity, and it has been found to be safe and to reduce the need for blood transfusions. EPO produced in the central nervous system7 is upregulated after insult and plays a role in neuroprotection. Experimental studies have reported that rhEPO possesses neuroprotective properties in different neonatal brain injury animal models, and clinical studies have shown that rhEPO treatment reduces brain injury and the incidence of neurological disabilities in infants.8,14-17 In addition, improved neurodevelopmental outcomes have been observed in preterm infants with anemia after rhEPO treatment. The neuroprotective effect of rhEPO was suggested to be through acting against apoptosis, inflammation, and neurotoxicity and by acting as an antioxidant in protecting white matter from injury and in promoting neural regeneration, injury repair, and normal development.

STUDY DESIGN Randomized, double-masked, placebo-controlled multicenter clinical trial. Research plan 400 infants will be randomized during the first three hours of life to receive EPO (5250 U/kg body weight) or placebo intravenously, the first dose(750U/kg) will be injected within 24h after birth, subsequent injection will be given each other day for 2 weeks. Standardized evaluation including cerebral sonography at day 1, 7 and 28 will determine the presence or absence of complications. Cerebral volume and white matter volume will be assessed at 40 postmenstrual weeks with MRI (only if available).

Experienced examiners will assess developmental function at 6 and 12 months corrected age using the reliable and validly revised Bayley Scales III of Infant Development and determine the presence or absence of impairment of motor function (cerebral palsy) and neurosensory function (blindness or deafness).

Primary outcome was cognitive development assessed with the Mental Development Index (MDI; norm, 100 [SD, 15]; higher values indicate better function) of the Bayley Scales of Infant Development, second edition (BSID-II) at 1 years corrected age.

Second outcome assess the effect of early administration of rh Epo on white matter development in preterm infants using Tract-based spatial statistics (TBSS ). White matter disease of the preterm infant, was semiquantitatively assessed from MRI at term-equivalent age based on an established scoring method.

ELIGIBILITY:
Inclusion Criteria:

* premature infants who admitted to the neonatal intensive care unit(NICU) Within 72 hours after birth, gestational ages younger than 32 weeks, birth weight less than 1500 gram, informed consent was obtained from the infants' parents or guardians

Exclusion Criteria:

* born with anemia, polycythemia, hemolysis and other hematological diseases
* hypertension,
* convulsions,
* a genetically defined syndrome
* a severe congenital malformation adversely affecting life expectancy or neurodevelopment
* severe intraventricular hemorrhage
* thrombosis disease
* other fatal diseases or which can seriously affect the prognosis

Max Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2017-04-10 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Neurodevelopmental outcome | corrected age of 18 months
  To evaluate neurodevelopmental function via Bayley Scales of Infant Development, second edition (BSID-II) at 18 months corrected age and gain incidence of MDI<70(Severe) or MDI<85(Moderate).

SECONDARY OUTCOMES:
TBSS（Tract-based spatial statistics） | corrected age of 40 weeks
  White matter disease of the preterm infant, was semiquantitatively assessed from MRI at term-equivalent age based on an established scoring method.

CONTACTS AND LOCATIONS:
Overall Officials: Xihui Zhou, Doctor, Principal Investigator — First Affiliated Hospital of Xian JiaotongUniversity
Locations (1):
- First Affiliated Hospital of Xian JiaotongUniversity, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] O'Gorman RL, Bucher HU, Held U, Koller BM, Huppi PS, Hagmann CF; Swiss EPO Neuroprotection Trial Group. Tract-based spatial statistics to assess the neuroprotective effect of early erythropoietin on white matter development in preterm infants. Brain. 2015 Feb;138(Pt 2):388-97. doi: 10.1093/brain/awu363. Epub 2014 Dec 22. PMID 25534356
- [Result] Wu YW, Mathur AM, Chang T, McKinstry RC, Mulkey SB, Mayock DE, Van Meurs KP, Rogers EE, Gonzalez FF, Comstock BA, Juul SE, Msall ME, Bonifacio SL, Glass HC, Massaro AN, Dong L, Tan KW, Heagerty PJ, Ballard RA. High-Dose Erythropoietin and Hypothermia for Hypoxic-Ischemic Encephalopathy: A Phase II Trial. Pediatrics. 2016 Jun;137(6):e20160191. doi: 10.1542/peds.2016-0191. Epub 2016 May 2. PMID 27244862
- [Result] Natalucci G, Latal B, Koller B, Ruegger C, Sick B, Held L, Bucher HU, Fauchere JC; Swiss EPO Neuroprotection Trial Group. Effect of Early Prophylactic High-Dose Recombinant Human Erythropoietin in Very Preterm Infants on Neurodevelopmental Outcome at 2 Years: A Randomized Clinical Trial. JAMA. 2016 May 17;315(19):2079-85. doi: 10.1001/jama.2016.5504. PMID 27187300
- [Result] Leuchter RH, Gui L, Poncet A, Hagmann C, Lodygensky GA, Martin E, Koller B, Darque A, Bucher HU, Huppi PS. Association between early administration of high-dose erythropoietin in preterm infants and brain MRI abnormality at term-equivalent age. JAMA. 2014 Aug 27;312(8):817-24. doi: 10.1001/jama.2014.9645. PMID 25157725
- [Result] Song J, Sun H, Xu F, Kang W, Gao L, Guo J, Zhang Y, Xia L, Wang X, Zhu C. Recombinant human erythropoietin improves neurological outcomes in very preterm infants. Ann Neurol. 2016 Jul;80(1):24-34. doi: 10.1002/ana.24677. Epub 2016 May 11. PMID 27130143